CLINICAL TRIAL: NCT05291221
Title: The Efficacy and Safety of Intratracheal Dexmedetomidine Versus Lidocaine for Smooth Tracheal Extubation in Patients Undergoing Eye-surgery.
Brief Title: Intratracheal Dexmedetomidine Versus Lidocaine in Eye Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, haidy salah mansour, Assistant professor in of Anesthesia and Intensive Care units in Minia University hospital, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22-2021
Record Dates: First submitted 2022-02-19; First posted 2022-03-22 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Postoperative Complications
Keywords: intratracheal; dexmedetomidine; eye-surgery; lidocaine
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control (Placebo Comparator): At the end of the operation by 15min, 5ml saline in a medical spray bottle was sprayed down the intratracheal tube of patients.
  Interventions: Drug: intratracheal saline
- Dexmedetomidine (Active Comparator): At the end of the operation by 15min, Dexmedetomidine (0.5µg/kg, diluted in 5mL saline in a medical spray bottle) was sprayed down the intratracheal tube of patients
  Interventions: Drug: intratracheal Dexmedetomidine
- Lidocaine (Active Comparator): At the end of the operation by 15min, (5ml) 2% of lidocaine was sprayed down the intratracheal tube of patients.
  Interventions: Drug: intratracheal Lidocaine

INTERVENTIONS:
Drug: intratracheal saline — At the end of the operation by 15min, 5ml of 0.9% normal saline was sprayed down the intratracheal tube of patients
  Other Names: Group C
  Arms: control
Drug: intratracheal Dexmedetomidine — At the end of the operation by 15min, Dexmedetomidine (0.5µg/kg, diluted in 5mL saline in a medical spray bottle) was sprayed down the intratracheal tube of patients
  Other Names: Group D
  Arms: Dexmedetomidine
Drug: intratracheal Lidocaine — At the end of the operation by 15min, (5ml) 2% of lidocaine was sprayed down the intratracheal tube of patients.
  Other Names: Group L
  Arms: Lidocaine

SUMMARY:
Cough during emergence from general anesthesia is considered a critical event as it may lead to surgical bleeding laryngospasm hemodynamic instability and could be life-threatening in patients who are at risk of complications related to increases in intracranial or intraocular pressure. Lidocaine administration has been widely used for reducing cough during extubation due to its simplicity and lack of serious adverse effects; There are two major routes for lidocaine administration systemic intravenous injection and local direct application on the laryngeal inlets such as spraying lidocaine on the supraglottic and subglottic regions or applying lidocaine jelly or sprayed. Dexmedetomidine is a potent alpha 2 selective adrenoceptor agonist and the most characteristic features include sympatholytic sedation analgesia and lack of respiratory depression. The aim of this study is to compare the effect of intratracheal dexmedetomidine and lidocaine on cough reflex in cataract surgery.

DETAILED DESCRIPTION:
The patients were randomly allocated into three groups each containing (40) patient. Group D received (0.5 μg/kg) of dexmedetomidine diluted and completed to 5 ml saline, Group L received (5ml) 2% of lidocaine and Group C received 5ml saline. The drugs were sprayed down the intratracheal tube of patients.

The following variables: Hemodynamic parameters HR, MAP, and SaO2 values in different times, preoperative IOP, cough, steward recovery score (SRS), detection of awareness and extubation time, the incidence of complications due to increasing IOP and surgeon satisfaction

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged from 18 to 60 years old
* ASA I or II class
* Undergo elective intraocular surgery
* Under general anesthesia.

Exclusion Criteria:

* Renal impairment
* Cardiorespiratory abnormalities
* Bronchial asthma COPD
* Restrictive lung diseases
* Liver failure
* Allergy to drugs will be used
* Patient refuse
* Pregnancy-lactation
* Significant obesity

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Cough reflex. | from time of awareness to 5 minute after extubation
  To evaluate efficacy and safety of both dexmedetomidine and lidocaine on Cough: from time of awareness to 5 minute after extubation 0= no cough
  1. minimal Cough (single)
  2. moderate cough<= 5S
  3. severe cough >=5S (bucking)

SECONDARY OUTCOMES:
mean arterial blood pressure | before anesthesia up to 30 minute after extubation
  Perioperative mean arterial blood pressure values were recorded
heart rate | before anesthesia up to 30 minute after extubation
  Perioperative heart rate values were recorded

CONTACTS AND LOCATIONS:
Overall Officials: Sohair A Magala, Lecturer, Study Director — Lecturer
Locations (1):
- Minya University, Minya, Egypt